CLINICAL TRIAL: NCT07085091
Title: A Phase 1, First in Human, Open-Label Multicenter Study to Evaluate ALX2004, an Antibody Drug Conjugate Targeting EGFR in Participants With Advanced or Metastatic Select Solid Tumors
Brief Title: A First in Human Study of ALX2004 With Advanced or Metastatic Selected Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ALX Oncology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ALX2004-01
Record Dates: First submitted 2025-06-27; First posted 2025-07-25 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: NSCLC (Advanced Non-small Cell Lung Cancer); HNSCC; CRC (Colorectal Cancer); ESCC; Colo-rectal Cancer; Head and Neck Cancer; Esophageal Squamous Cell Carcinoma (ESCC)
Keywords: ALX2004; EGFR; Solid Tumors; metastatic; Antibody Drug Conjugate; ADC; HNSCC; CRC; Lung; Non small cell lung cancer; esophageal; EGFR ADC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Colorectal Neoplasms; Colonic Neoplasms; Head and Neck Neoplasms; Esophageal Squamous Cell Carcinoma; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: The dose escalation and dose exploration portions of the study will be non-randomized. For each tumor type selected for dose expansion, either one or two dose(s) and schedule(s) may be tested. If two doses/schedules are tested, allocation will be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ALX2004 Phase 1a (Dose Escalation) (Experimental): ALX2004 will be administered. Patients will be enrolled into escalating dose levels during the dose escalation phase
  Interventions: Drug: ALX2004
- ALX2004 Phase 1a (Dose Exploration) (Experimental): ALX2004 will be administered. All or a subset of tumors tested in dose escalation will enroll into 1 or 2 dose levels during the dose exploration phase
  Interventions: Drug: ALX2004
- ALX2004 Phase 1b (Dose Expansion) (Experimental): ALX2004 will be administered. Patients will receive the recommended phase 2 dose during the dose expansion phase
  Interventions: Drug: ALX2004

INTERVENTIONS:
Drug: ALX2004 — ALX2004 is a novel ADC targeting EGFR. Drug: ALX2004 IV Infusion
  Arms: ALX2004 Phase 1a (Dose Escalation)
Drug: ALX2004 — ALX2004 is a novel ADC targeting EGFR. Drug: ALX2004 IV infusion
  Arms: ALX2004 Phase 1a (Dose Exploration)
Drug: ALX2004 — ALX2004 is a novel ADC targeting EGFR. Drug: ALX2004 IV infusion
  Arms: ALX2004 Phase 1b (Dose Expansion)

SUMMARY:
A Phase 1, First in Human, Open-Label Multicenter Study to Evaluate ALX2004, an Antibody Drug Conjugate Targeting EGFR in Participants with Advanced or Metastatic Select Solid Tumors

DETAILED DESCRIPTION:
This study consists of Phase 1a Dose finding, comprising of Dose Escalation portion followed by Dose Exploration, and a Phase 1b Dose Expansion. The study will enroll previously treated advanced or metastatic non-small cell lung cancer (NSCLC), head and neck squamous cell carcinoma (HNSCC), esophageal squamous cell carcinoma (ESCC) and colorectal cancer (CRC). Up to 170 patients are expected to be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with locally advanced, recurrent or metastatic histologically confirmed HNSCC, NSCLC, ESCC, CRC (left sided); locally advanced or recurrent disease must not be amenable to resection with curative intent

  1. Dose Escalation: Participants who have relapsed or progressed following prior anticancer therapy in the advanced/metastatic setting and for whom no approved or standard therapy is available.
  2. Dose Exploration and Dose Expansion: The following tumor-specific criteria also apply. These cohorts will include all or a subset of these tumors.

HNSCC - Received no more than 3 prior lines of therapy in the advanced or metastatic setting

NSCLC - For participants with a targetable molecular alteration: received appropriate standard targeted therapy and no more than 2 prior lines of systemic chemotherapy in the advanced/metastatic setting. For participants without a targetable molecular alteration: received platinum-based chemotherapy and CPI (in combination or separately), and have received no more than 2 prior lines of systemic chemotherapy in the advanced/metastatic setting

ESCC - Received no more than 3 prior lines of therapy in the advanced/metastatic setting

CRC (left-sided) - For participants with a targetable molecular alteration (including dMMR or MSI-H): Received appropriate standard therapy for the alteration, at least 2 prior lines of systemic chemotherapy, and no more than 4 prior lines of therapy in the advanced/metastatic setting. For participants without a targetable molecule alteration: Received at least 2 prior lines of systemic chemotherapy (including an oxaliplatin-based chemotherapy), vascular endothelial growth factor (VEGF)-based therapy, and no more than 4 prior lines of therapy in the advanced/metastatic setting.

* Adequate Bone Marrow Function
* Adequate Renal & Liver Function
* Adequate Performance Status

Exclusion Criteria:

* Participants with disease suitable for local therapy with curative intent.
* Has a life expectancy of less than 3 months and/or has rapidly progressing disease (e.g., tumor bleeding, uncontrolled tumor pain) in the opinion of the treating investigator
* Prior treatment with any ADCs that have an active TOP1 inhibitor-based component

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Incidence of dose limiting toxicities (DLTs) | Up to 28 days
  Phase 1a: Number and proportion of participants enrolled in the dose escalation phase who experience dose-limiting toxicities (DLTs), received at least one dose of ALX2004 and completed the DLT evaluation
Phase 1a: Incidence of treatment emergent adverse events | Up to 2 years from first dose
  Phase 1a: Adverse Events as characterized by type, frequency, severity (NCI CTCAE v5.0), timing, seriousness, and relationship to the study drug in order to establish the RDE. Laboratory abnormalities as characterized by type, frequency, severity and timing
Phase 1b: Overall Response Rate (ORR) per investigator assessment using RECIST v1.1 | Up to 2 years from first patient dosed in dose expansion phase
  Phase 1b: ORR is defined as proportion of participants whose BOR is complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
Phase 1a and 1b: Maximum Concentration (Cmax) | Up to 2 years
  To evaluate the Cmax of ALX2004
Phase 1a and 1b: Time of Maximum Plasma Concentration (Tmax) | Up to 2 years
  To evaluate the Tmax of ALX2004
Phase 1a and 1b: Clearance (CL) | Up to 2 years
  To evaluate the clearance of ALX2004
Phase 1a and 1b: Area under the concentration time curve (AUC) | Up to 2 years
  To evaluate the AUC of ALX2004
Phase 1a and 1b: Terminal elimination half-life (t1/2) | Up to 2 years
  To evaluate the t1/2 of ALX2004
Phase 1a: Overall Response Rate (ORR) per investigator assessment using RECIST v1.1 | Up to 2 years from first dose
  Phase 1a: ORR is defined as proportion of participants whose BOR is complete response (CR) or partial response (PR)
Phase 1a and 1b: Evaluate the immunogenicity of ALX2004 | Phase 1a: Up to 2 years from first dose. Phase 1b: Up to 2 years from first patient dosed in dose expansion phase
  Measured by the presence of human plasma ADA (Anti-ALX2004 antibodies)
Phase 1b: Incidence of treatment emergent adverse events | Up to 2 years from first patient dosed in dose expansion phase
  AEs as characterized by type, frequency, severity (as graded by the NCI CTCAE v.5.0) timing, seriousness, and relationship to study drug. Laboratory abnormalities as characterized by type, frequency, severity and timing
Phase 1a and 1b: Progression Free Survival (PFS) | Phase 1a: Up to 2 years from first dose. Phase 1b: Up to 2 years from first patient dosed in dose expansion phase
  PFS is defined as the time (in months) from the date of the first dose of ALX2004 to the date of the first instance of progressive disease or death
Phase 1a and 1b: Overall Survival (OS) | Phase 1a: Up to 2 years from first dose. Phase 1b: Up to 2 years from first patient dosed in dose expansion phase
  OS is defined as the time (in months) from the date of the first dose of ALX2004 to the date of death
Phase 1a and 1b: Best Overall Response (BOR) | Phase 1a: Up to 2 years from first dose. Phase 1b: Up to 2 years from first patient dosed in dose expansion phase
  BOR is defined as the best response reached during the course of the trial from the response categories of CR, PR, SD, PD, and No Response using RECIST v1.1
Phase 1a and 1b: DCR (Disease Control Rate) | Phase 1a: Up to 2 years from first dose. Phase 1b: Up to 2 years from first patient dosed in dose expansion phase
  DCR is defined as the proportion of participants whose BOR is PR, CR, or SD
Phase 1a and 1b: Duration of Response (DoR) | Phase 1a: Up to 2 years from first dose. Phase 1b: Up to 2 years from first patient dosed in dose expansion phase
  DoR is defined as the time (in months) from the first instance of a BOR, of CR/PR until the date of the first instance of progressive disease

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - ALX Center 3, Grand Rapids, Michigan
  - ALX Center 6, Portland, Oregon
  - ALX Center 5, Houston, Texas
  - ALX Center 4, West Valley City, Utah
  - ALX Center 2, Fairfax, Virginia
  - ALX Center 1, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No